CLINICAL TRIAL: NCT05503446
Title: Using Commonly Available Food Products To Treat Food Allergy (NATASHA Study)
Brief Title: Using Commonly Available Food Products To Treat Food Allergy
Acronym: NATASHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Imperial College London (Other); Natasha Allergy Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERGO 71012; IRAS ID 310316 (Other: NHS Human Research Authority)
Record Dates: First submitted 2022-07-06; First posted 2022-08-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: IgE-Mediated Cow Milk Allergy; Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Parallel arm, with cross-over for those allocated to control group only following determination of primary outcome
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessed by double-blind, placebo-controlled food challenge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Immunotherapy, in-hospital supervision for updosing (Experimental): Active oral immunotherapy, with all updosing visits taking place in hospital
  Interventions: Other: Peanut in common foods or supermarket-sourced cow's milk (CM)
- Oral Immunotherapy, virtual supervision for updosing (Experimental): Active oral immunotherapy, with all updosing visits taking place with virtual supervision
  Interventions: Other: Peanut in common foods or supermarket-sourced cow's milk (CM)
- Control arm: allergen avoidance (No Intervention)

INTERVENTIONS:
Other: Peanut in common foods or supermarket-sourced cow's milk (CM) — Participants will be given a set dose of peanut (e.g. peanut-containing cereal, whole peanuts) or cow's milk to take on a daily basis, as per protocol
  Arms: Oral Immunotherapy, in-hospital supervision for updosing; Oral Immunotherapy, virtual supervision for updosing

SUMMARY:
Food allergy affects 1 in 30 children, and is the commonest trigger for life-threatening reactions (anaphylaxis) in this age group. It is a major public health issue, with practical implications for industry, education and healthcare systems. Oral immunotherapy (OIT) is an emerging treatment option, where small, increasing doses of a food allergen are used to cause "desensitisation", so food-allergic individuals no longer have symptoms when exposed to the trigger food. However, frequent allergic reactions during OIT (including anaphylaxis) are common, and can lead to patients having to stop treatment. In addition, food-allergic children usually dislike the taste of the food they are allergic too, which affects compliance and treatment success. There is a lack of longer-term data to inform cost-effectiveness analyses for OIT.

The NATASHA study will recruit young people from age 6+ years with IgE-mediated peanut allergy, and young people aged 3+ years with IgE-mediated allergy to cow's milk, who will undergo oral immunotherapy for these allergens using real-world foods (taken carefully according to a standardised protocol under medical supervision). In addition to assessing efficacy and safety outcomes, we will also collect longer-term data to evaluate cost-effectiveness in the UK setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-23 years with IgE-mediated peanut allergy, or age 3-23 years with IgE-mediated food allergy to cow's milk
2. Past history consistent with IgE-mediated allergy to the relevant allergen
3. Allergic to cumulative ≤1.44 g protein (of the specific allergen) at baseline DBPCFC, prior to treatment allocation
4. Written informed consent (for young people under 16, consent from the parent/legal guardian (AND assent from the young person when the young person is age 6+ years)

Exclusion Criteria:

1. Required previous admission to an intensive care unit for management of an allergic reaction
2. Clinically significant chronic illness (other than asthma, rhinitis or eczema)
3. Moderate-severe eczema, defined as requiring more than once daily application of 1% hydrocortisone or equivalent topical calcineurin inhibitor as maintenance treatment despite appropriate use of emollients (eczema is not otherwise an exclusion criteria)
4. Poorly controlled asthma within the previous 3 months (as defined by clinician judgement with reference to the International Consensus On (ICON) Pediatric Asthma consensus), or asthma requiring treatment with >5 days oral corticosteroids within the previous 3 months
5. Previous history of eosinophilic oesophagitis
6. Undergoing subcutaneous or sublingual immunotherapy to respiratory allergens, and not yet established on maintenance dosing for at least 6 months
7. Undergoing allergen immunotherapy for food allergy and within the first year of treatment
8. In CM-allergic children under consideration for desensitisation to CM:

   * currently consuming CM-containing products other than extensively-heated milk in baked foods (e.g. biscuits, cakes)
   * significant symptoms of non-IgE-mediated CM allergy within the previous 12 months
9. Taking prebiotic or probiotic supplements and unwillingness to discontinue
10. Subjects receiving anti-IgE therapy, oral immunosuppressants, beta-blocker or Angiotensin Converting Enzyme (ACE) inhibitor
11. Tolerance to cumulative ≥1.44 g food protein at initial DBPCFC during screening
12. Objective allergic reaction to ≤4mg cow's milk protein or ½ Reese's puff in peanut-allergic children, during screening
13. Objective reaction to the placebo at screening DBPCFC
14. Past or current medical issue, participation in another clinical trial or other consideration, which, in the opinion of the investigator, may pose additional risks from study participation, interfere with compliance or otherwise impact on the quality or interpretation of study data
15. Pregnancy
16. Direct personal or commercial relationship with a member of the local study team directly involved with the conduct of the trial
17. Unwilling or unable to fulfil study requirements, including the requirement for appropriate supervision following dosing at home)

Ages: 3 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and effectiveness | 9-12 months
  The proportion of participants in intervention arms (combined) versus control arm (by allergen) who, following 9-12 months of OIT (or standard care, for controls):
  * tolerate at least 1 gram of food protein (discrete dose, approximately 4-6 peanuts, or 30ml of CM) AND
  * demonstrate a minimum 10-fold increase in the maximum tolerated dose (defined as the highest dose not causing dose-limiting symptoms) at the end-of-updosing double-blind, placebo-controlled food challenge (DBPCFC), compared to baseline DBPCFC

SECONDARY OUTCOMES:
Safety: adverse events | 24 months
  i. Proportion of participants experiencing study-related adverse events (excluding mild, transient oropharyngeal symptoms) in active vs control arms, by allergen ii. Other safety outcomes: rate of anaphylaxis (and adrenaline [epinephrine] use), withdrawals due to intervention, by allergen iii. Adverse events (excluding mild, transient oropharyngeal symptoms) specifically occurring at updosing visits, in the home versus in-hospital updosing groups, by allergen
Health-related quality of life (HRQL) as assessed by the Food Allergy Quality of Life Questionnaire (FAQLQ) | 24 months
  Change in HRQL score assessed using validated questionnaire (Food Allergy Quality of Life Questionnaires (FAQLQ), from baseline at the following timepoints post allocation: 3, 6, end of induction (9-12 months), 18 and 24 months, in i. Participants ii. Parent/carers (if participants aged ≤17 years)
  The tools to be used are:
  - FAQLQ: as per Muraro et al, Allergy 2014; 69:845-853. A higher score is associated with a greater impact on quality of life, as per the cited reference.
Health-related quality of life (HRQL) as assessed by EQ5D | 24 months
  Change in quality of life assessment assessed using EQ5D, from baseline at the following timepoints post allocation: 3, 6, end of induction (9-12 months), 18 and 24 months, in i. Participants ii. Parent/carers (if participants aged ≤17 years)
  The tools to be used are:
  - EQ5D: a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys (see https://euroqol.org/ for detailed instructions on use)
Health-related quality of life (HRQL) as CHU9D | 24 months
  Change in quality of life assessment assessed using CHU9D, from baseline at the following timepoints post allocation: 3, 6, end of induction (9-12 months), 18 and 24 months, in i. Participants ii. Parent/carers (if participants aged ≤17 years)
  The tools to be used are:
  - CHU9D - a paediatric generic preference-based measure of health-related quality of life suitable for 7 to 17 year olds. (see https://licensing.sheffield.ac.uk/product/CHU-9D for detailed instructions on use)
Adherence to dietary avoidance | 24 months
  Adherence to dietary avoidance between intervention and control arms (by allergen, and between allergens) as determined by number of accidental reactions reported by each participant, during the duration of the study
Adherence to treatment | 24 months
  Adherence to daily OIT dosing by allergen, expressed as a the proportion of doses taken divided by the number of doses which should have been taken by each participant.
Immunological outcomes: change in skin prick test wheal | 24 months
  Change in immunological measures (skin prick test wheal (mm diameter) to commercial allergen extract, performed according to national guidelines) at baseline vs 12 months vs 24 months, between active and control arms (by allergen)
Immunological outcomes: change in allergen-specific serum antibody profile | 24 months
  Change in immunological measures (specific Immunoglobulin E (IgE) to specific allergen) measured by ImmunoCAP (kUA/l) at baseline vs 12 months vs 24 months, between active and control arms (by allergen)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, FRCPCH PhD, Principal Investigator — Imperial College London
Locations (5):
- United Kingdom (5):
  - University of Hospitals of Leicester NHS Trust, Leicester
  - Imperial College Healthcare NHS Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Sheffield Children's Hospital NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No
Deidentified data may be available upon request to the Chief Investigators, subject to local data protection legislation.